CLINICAL TRIAL: NCT00204633
Title: Randomized Phase II-Trial to Determine the Impact of Darbepoetin Alfa on the Frequency of RBC Transfusions in Patients With Metastatic "Poor Prognosis" Germ Cell Tumor Treated With High-Dose Chemotherapy (HD-VIP Regimen)
Brief Title: Darbepoetin Alfa in Patients With "Poor Prognosis" Germ Cell Tumor Treated With High-Dose Chemotherapy (HD-VIP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jth_004
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Dysgerminoma
MeSH Terms: conditions — Dysgerminoma | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa

SUMMARY:
The aim is to determine the frequency of RBC transfusion in patients with metastatic "poor prognosis" germ cell tumor during high-dose chemotherapy (HD-VIP, level 6) with or without Darbepoetin alfa

ELIGIBILITY:
Inclusion Criteria:

* Poor prognosis" according IGCCCG-criteria:
* Primary mediastinal tumor
* Gonadal/retroperitoneal germ cell tumor with visceral metastases except of lung
* Poor marker: AFP > 10.000 ng/ml or beta-HCG > 10.000 ng/ml (50.000 IU/l) andd LDH >10 x upper normal limit
* No previous chemotherapy
* Age > 18 years
* Performance-Status: WHO =< 2
* Written informed consent
* Ability to give informed consent

Exclusion Criteria:

* Hemolysis
* Hematological disease with insufficient erythropoiesis
* Patients without sufficient treatment of sideropenia, folate deficiency or vitamin B12 deficiency
* Uncontrolled arterial hypertension
* Treatment with rh-Erythropoetin during trial
* Creatinin clearance < 50 ml/min
* Insufficient bone marrow function (WBC count < 3.000/ml or platelets < 100.000/µl)
* Other major symptomatic or uncontrolled illnesses not allowing to complete treatment protocol with the exception of symptoms caused by the primary disease
* Second malignancy, except of completely resected basal cell carcinoma of the skin

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2003-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
frequency of transfusions (reduction from 90% to 65%)

SECONDARY OUTCOMES:
proportion of patients with no transfusions
developing of hemoglobin levels
objective remission rate
progression-free- and overall-survival (pfs, os)
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Joerg T. Hartmann, MD, Principal Investigator — South West German Cancer Center, Medical Center II, University of Tuebingen
Locations (1):
- Medical Center II, University of Tuebingen, Tübingen, Germany